CLINICAL TRIAL: NCT05866757
Title: Discontinuation of Maintenance Therapy for the Patients Diagnosed With Multiple Myeloma in Sustainable Minimal Residual Disease (MRD) Negative Remission Without High Risk Features
Brief Title: Discontinuation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Cancer Research@UCC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22107
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma; Cancer; Hematologic Cancer
Keywords: Multiple Myeloma; Cancer
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be divided in the following groups:
  Group 1: Patients with biochemically detectable disease who have failed to achieve Complete remission (CR) or Very good Partial Remission (VGPR) by IMWG criteria and/or MRD-positive and/or high risk features. They will continue maintenance therapy until disease progression with monitoring every 3 months as per standard of care (SOC), or more often if required.
  Group 2: Patients in biochemical remission, who meet IMWG criteria for very good partial response (VGPR) or complete response (CR and and sustained MRD (defined as MRD-negative at two time points that are at least 1 year apart) without high risk features This group will be divided in the following subgroups:
  Subgroup A: Patients who prefer to continue on maintenance therapy. Maintenance will continue until disease progression.
  Subgroup B: Patients who prefer to discontinue maintenance therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continuation - Group 1: Detectable disease (No Intervention): Continuing Maintenance Therapy- Patients with biochemically detectable disease who have failed to achieve Complete remission (CR) or Very good Partial Remission (VGPR) by IMWG criteria and/or MRD-positive and/or high risk features. They will continue maintenance therapy until disease progression with monitoring every 3 months as per standard of care (SOC), or more often if required. In case of disease progression these patients will be switched to a different treatment and withdraw from the study. QOL will be assessed.
- Continuation - Group 2 Subgroup A: Remission (No Intervention): Continuing Maintenance Therapy- Patients in biochemical remission, who meet IMWG criteria for very good partial response (VGPR) or complete response (CR and and sustained MRD (defined as MRD-negative at two time points that are at least 1 year apart) without high risk features. High-risk cytogenetics abnormalities defined as per IMWG criteria (del(17p) and/or t(4;14) and/or t(14;16)) , or any other features suggestive of high risk disease: extramedullary disease, poor response to first line therapy, plasma cell leukaemia, organomegaly secondary to infiltration by multiple myeloma.
  Maintenance will continue until disease progression, monitored every 3 months as per SOC or more often if required. In case of disease progression these patients will be switched to a different treatment and withdraw from the study. QOL will be assessed.
- Discontinuation - Group 2 Subgroup B (Other): Patients who prefer to discontinue maintenance therapy. Patients who have discontinued maintenance therapy earlier than 2 years due to side effects but also achieved sustained MRD negative CR might be also included in this subgroup. This subgroup will be monitored and per SOC with blood tests, and BM MRD by NGF. In case of detectable disease in any of the samples (blood or BM) they will be offered to restart on maintenance therapy. Changing to a different type of treatment could be also offered to these patients, after discussion with treating physician. In case of being switched to a different treatment patient will withdraw from the study. QOL will be assessed
  Interventions: Other: Discontinuation of maintenance treatment

INTERVENTIONS:
Other: Discontinuation of maintenance treatment — The discontinuation of maintenance treatment in multiple myeloma. Classed as interventional due to treatment being taken away.
  Arms: Discontinuation - Group 2 Subgroup B

SUMMARY:
An interventional, non-randomised study to assess the risk of progression after discontinuation of maintenance therapy in sustained MRD negative complete remission by flow cytometry MM patients without high-risk features who have completed at least two years of maintenance therapy or who have discontinued maintenance due to side effects. The primary endpoint is to assess the rates of sustained MRD negativity by NGF in the bone marrow at 12 months after discontinuation of maintenance therapy.

DETAILED DESCRIPTION:
Up to 70 patients over 18 years of age who have a diagnosis of Multiple Myeloma and have completed at least 2 years of maintenance therapy.

Participants would be divided in two groups: Group 1. Patients with detectable disease who have not achieved CR or VGPR as per IMWG criteria and/or detectable MRD and/or high risk features detectable disease, failed to achieve Complete Remission (CR) or Very Good Partial Remission (VGPR) continuing on maintenance therapy. Group 2. Patients who meet International Myeloma working Group (IMWG) criteria for very good partial response (VGPR) or complete response (CR). Patients who have achieved sustained MRD negative remission by next generation flow cytometry (NGF),defined by IMWG as MRD-negative at two time points that are at least 1 year apart, To the participants in this group will be offered to discontinue maintenance therapy, and it will be further divided in the following subgroups: Subgroup A) Patients who are willing to continue maintenance therapy. Subgroup B) Patients who are willing to discontinue maintenance therapy and continue monitoring. This subgroup will also include patients who have discontinued maintenance therapy earlier than 2 years due to side effects but also achieved sustained MRD negative CR might be also included.

The number of the study participants will be limited by the number of patients treated in Cork University Hospital who are meeting inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or over
2. Patient with diagnosis of multiple myeloma as per IMWC in first line of treatment (induction, consolidation, ASCT, maintenance is considered single line therapy for the purpose of this study, also discontinuation of 1 maintenance regimen due to toxicity and start of another is considered single line therapy for the purpose of this study).
3. Received at least 2 years of maintenance therapy, defined as any anti-myeloma therapy to prevent disease recurrence and prolong time in remission
4. Patients who have discontinued maintenance therapy earlier than 2 years due to side effects but also achieved sustained MRD negative CR might be also included
5. Patients must be able to understand and be willing to sign a voluntary informed consent form and agree to compliance with the protocol schedule, with the knowledge that they may withdraw consent at any time without impact on future medical care.

Exclusion Criteria:

1. Patients who have received more than one line of therapy (induction, consolidation, ASCT, maintenance is considered single line therapy for the purpose of this study, also discontinuation of 1 maintenance regimen due to toxicity and start of another is considered single line therapy for the purpose of this study) or patients who have not completer two years of maintenance therapy, unless maintenance was discontinued voluntarily and the patient has achieved sustainable MRD negative remission..
2. Patients with plasma cell disorders other than MM: lymphoplasmacytic lymphoma/Waldenstrom macroglobulinemia, AL amyloidosis, POEMS syndrome (Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, and Skin changes), etc…
3. Prior organ transplant or condition requiring immunosuppressive therapy.
4. Prior allogenic haematopoietic cell transplant
5. Treatment with any investigational therapy that does not include maintenance as a part of the treatment strategy.
6. Unable to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants that remain in sustained MRD negative remission by NGF in the bone marrow at 12 months after discontinuation of maintenance therapy. | 12 months
  Number

SECONDARY OUTCOMES:
Number of participants that remain in sustained MRD negative remission by NGF in the bone marrow at 24 months after discontinuation of maintenance therapy. | 24 months
  Number
Progression-free survival in multiple myeloma patients at 1 year in both groups of patients (on maintenance therapy and those who have discontinued) | 1 year
  Number
Progression-free survival in multiple myeloma patients at 2 years in both groups of patients (on maintenance therapy and those who have discontinued) | 2 years
  Number
Compare health-related quality of life between MM patients discontinuing versus continuing maintenance therapy using a QOL questionnaire. The EoRTC QLQ - MY20 will be used. Minimum value 50, maximum value 200. Lower values indicate better outcomes. | 2 years
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Ireland, Ireland